CLINICAL TRIAL: NCT01653522
Title: The Impact of Triptan and Doxycycline on Neuroinflammatory Biomarkers in Acute Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-061
Record Dates: First submitted 2012-07-23; First posted 2012-07-31 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Migraine Disorders; Headache, Migraine; Migraine; Migraine Headache; Migraine With Aura; Migraine Without Aura; Headache Disorders, Primary
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache Disorders, Primary | interventions — Tryptamines; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Triptan (Experimental)
  Interventions: Drug: Triptan
- Doxycycline (Experimental)
  Interventions: Drug: Doxycycline
- Triptan + Doxycycline (Experimental)
  Interventions: Drug: Triptan; Drug: Doxycycline
- Control (No Intervention)

INTERVENTIONS:
Drug: Triptan
  Arms: Triptan; Triptan + Doxycycline
Drug: Doxycycline
  Arms: Doxycycline; Triptan + Doxycycline

SUMMARY:
The purpose of this study is to determine the effects of triptans and doxycycline on neuroinflammatory markers in acute migraine.

DETAILED DESCRIPTION:
Increased inflammatory cytokines and matrix metalloproteinases (MMPs) have been recently implicated in migraine. Inflammation may be a key player in the pathophysiology of migraine by altering blood-brain barrier (BBB) function. As an inflammation induced MMP, MMP-9 is involved in both BBB disruption and neuropathic pain, and is largely derived by neutrophil degranulation during neutrophil-BBB interaction. The tetracycline group of antibiotics may suppress MMP production and neutrophil degranulation. This study aims to investigate known neuroinflammatory biomarkers with a focus on BBB breakdown during acute migraine attacks and assess marker responses to conventional treatment (triptans) and novel MMP targeted therapy (doxycycline). This pilot project data will supplement future projects investigating novel therapeutic strategies such as MMP inhibitors in both migraine acute treatment and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of migraine with or without aura that fulfill the 2nd Edition of The International Headache Classification (ICHD-II) criteria
* Active prescription for an oral triptan medication to abort acute migraines

Exclusion Criteria:

* Tetracycline group or other anti-inflammatory medication use in the preceding three months
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Serum neuroinflammatory marker concentrations

SECONDARY OUTCOMES:
Headache intensity (four-point scale)
Number of participants with adverse events as a measure of safety and tolerability
Time to headache relief
Time to headache recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen E Lakhan, MD, PhD, MEd, MS, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No